CLINICAL TRIAL: NCT04824105
Title: Modeling and Modulating Mechanisms of Escape, Avoidance, and Approach in the Anxiety Disorder Spectrum
Brief Title: Modulating Anxious Coping
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 00106843; 1K23MH123931-01A1 (NIH)
Record Dates: First submitted 2021-03-24; First posted 2021-04-01 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Anxiety Disorders
MeSH Terms: conditions — Anxiety Disorders | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neurostimulation Group (Experimental): On one study day, participants will complete experimental tasks during functional magnetic resonance imaging. On two other study days, participants will complete tasks before and after receiving repetitive transcranial magnetic stimulation (rTMS). All participants will receive rTMS to ventromedial prefrontal cortex on one study day, and to pre-supplementary motor area on another study day.
  Two stimulation procedures will be used, one for ventromedial prefrontal cortex and one for pre-supplementary motor area. For both targets, 3 sessions of 600 pulses at 110% of resting motor threshold will be presented over 30 minutes. For ventromedial cortex, a session will involve intermittent theta burst triplets at 50 Hz for 2 seconds and repeated every 10 seconds for a total of 190 seconds. For pre-supplementary motor area, a session will involve continuous theta burst presented in 3-pulse bursts with 15 pulses/ sec.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS)

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation (rTMS) — A repetitive Transcranial Magnetic Stimulation (rTMS) MagVenture MagPro TMS System will be used to deliver intermittent theta burst to ventromedial prefrontal cortex, and continuous theta burst to pre-supplementary motor area.

SUMMARY:
This is a study to find out if a device that temporarily alters brain activity (repetitive transcranial magnetic stimulation, rTMS) might be used to change how people with anxiety or related concerns cope with feared or anxiety-producing situations. The study is recruiting people who recently started treatment for anxiety or a related concern. The study involves 3 visits to the Medical University of South Carolina. At the first visit, participants do interviews and surveys asking about anxiety and related concerns, and they also do tasks where they see and react to emotional pictures while their brain activation is measured. At the next two visits, participants receive rTMS, which works by rapidly turning a focused magnetic field on and off repeatedly over the head in a way that passes directly through the hair, scalp, and skull and onto the brain and can temporarily increase brain activity under the magnetic field. After rTMS, participants do two tasks where they see and react to emotional situations while wearing sensors on their hand, arms, face, and head.

Each visit in this study is expected to last between 2 - 4 hours. This is not a treatment study, but the study is being conducted with the hope that it will help improve treatment in the future.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 65 y.o.
* Meets criteria for an anxiety disorder (Generalized Anxiety Disorder, Panic Disorder, Social Anxiety Disorder, Specific Phobia), posttraumatic stress disorder, obsessive- compulsive disorder, or current adjustment disorder with anxiety
* Is currently seeking mental health treatment
* Is able to read consent document and provide informed consent.
* English is a first or primary fluent language.

Exclusion Criteria:

* Current alcohol or substance use disorder of more than mild severity (as defined by DSM-5 and determined using standardized self-report instruments)
* Lifetime diagnosis of psychotic disorder or bipolar mania
* Presence of neurological disorder that contraindicates TMS or neurophysiological recording: Seizure disorder Lifetime history of traumatic brain injury with loss of consciousness Neurodegenerative disorder (e.g., Alzheimer's Disease, Parkinson's Disease, Frontotemporal Dementia)
* Presence of other medical disorder that would make it too uncomfortable to sit or lie still for long recording periods
* Presence of standard contraindications for MRI or rTMS Metal in the body Currently pregnant Claustrophobia Significant sensitivity to noise Medical conditions or treatments that lower seizure threshold History of severe brain injury History of seizures/ epilepsy
* Currently taking anticholinergic mediation, neuroleptic medication, or sedative/ hypnotic medication Note: SSRI, cholinesterase inhibitors or NMDA receptor antagonists are allowed if patient has been on a stable regimen of four weeks prior to enrollment
* Currently taking chronic opiate medications or substances
* Currently taking naltrexone

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-06-26 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Fear-Potentiated Startle Reflex | Immediately Pre-Stimulation and Immediately Post-Stimulation (Approx. 30 minutes between assessments)
  Fear-potentiated startle is measured during an experimental task in which participants prepare to avoid, escape, or simply be exposed to aversive pictures. Fear-potentiated startle measures motivational activation during the preparation period.
Change in Speed to Initiate Avoidance Behavior | Immediately Pre-Stimulation and Immediately Post-Stimulation (Approx. 30 minutes between assessments)
  Reaction time to initiate flight is measured in an experimental task in which participants can win money but also must evade a slow, moderate, or fast virtual predator. Reaction time measures behavioral tendency to approach or avoid.

SECONDARY OUTCOMES:
Change in Escape/ Avoidance Electroencephalography | Immediately Pre-Stimulation and Immediately Post-Stimulation (Approx. 30 minutes between assessments)
  Electroencephalography (EEG) is measured during an experimental task in which participants prepare to avoid, escape, or simply be exposed to aversive pictures. An event-related potential, the stimulus-preceding negativity, will be derived from the EEG to index action preparation processing.
Change in Approach/ Avoidance Conflict Electroencephalography | Immediately Pre-Stimulation and Immediately Post-Stimulation (Approx. 30 minutes between assessments)
  Electroencephalography (EEG) is measured during an experimental task in which participants can win money but also must evade a slow, moderate, or fast virtual predator. A frequency signature, power in the theta frequency band, will be derived from the EEG to index cognitive control processes.
Change in Task-Related Heart Rate Changes | Immediately Pre-Stimulation and Immediately Post-Stimulation (Approx. 30 minutes between assessments)
  Heart rate is measured during experimental tasks in which: 1) participants prepare to avoid, escape, or simply be exposed to aversive pictures; 2) participants can win money but also must evade a slow, moderate, or fast virtual predator. Heart rate slowing measures task-related engagement of attention, while heart rate increase indicates defensive activation.
Change in Task-Related Skin Conductance Responding | Immediately Pre-Stimulation and Immediately Post-Stimulation (Approx. 30 minutes between assessments)
  Skin conductance is measured during experimental tasks in which: 1) participants prepare to avoid, escape, or simply be exposed to aversive pictures; 2) participants can win money but also must evade a slow, moderate, or fast virtual predator. Skin conductance increases indicate task-related sympathetic arousal.
Change in Task-Related Perceived Control | Immediately Pre-Stimulation and Immediately Post-Stimulation (Approx. 30 minutes between assessments)
  Perceived control over aversive stimuli is queried after an experimental task in which participants prepare to avoid, escape, or simply be exposed to aversive pictures. Perceived control for each condition is queried using self-report Likert-type scales for each condition.
Change in Difficulty of Avoiding Task-Based Aversive Exposure | Immediately Pre-Stimulation and Immediately Post-Stimulation (Approx. 30 minutes between assessments)
  Difficulty of avoiding exposure to aversive stimulation is queried after each trial during a task in which participants can win money but also must evade a slow, moderate, or fast virtual predator. Avoidance difficulty is queried using a Likert-type scale delivered after each trial. The scale ranges from 1 to 5, with higher scores indicating greater perceived difficulty of avoiding capture by the virtual predator.
Change in State Anxiety During Session | Immediately Pre-Stimulation and Immediately Post-Stimulation (Approx. 30 minutes between assessments)
  State-level anxiety is measured throughout the experimental session using the State-Trait Anxiety Inventory - State Form. The State-Trait Anxiety Inventory - State Form uses 20 items querying anxiety symptom experience in the present moment to measure how anxiety fluctuates across the experimental session. The scale ranges from 20 to 80, with higher scores indicating higher state anxiety.

OTHER OUTCOMES:
Task-Related Brain Activation | During Session (Approx. 45 minutes)
  Blood flow in the brain will be measured during completion of two experimental tasks using functional magnetic resonance imaging (fMRI). Blood flow in the brain can be used to measure what brain areas are being activated during the performance of a task.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Objective data will be archived in raw format on the NITRIC Data Repository. Sufficient description of tasks and event markers will be included to allow reprocessing and replication by trained researchers. Original, albeit cleaned and de-identified, self-report data will also be included. Cleaning will entail the most basic review of each variable to assure correct coding, and, in justified cases, invert variable scores to make variables easier to interpret. Inversions will always be noted.
  DATA FORMAT: Objective data will be delivered to NITRIC in NIFTII format for fMRI data and tab-delimited text files for EEG and physiology data. Self-report data will be delivered in SPSS .sav format. No identifying information will be included.
  VARIABLE CREATION: All variable computation, weighting, and imputation syntax will be in SPSS format and delivered in .txt file. A variable definition list / codebook will also be delivered.
Supporting Information: Study Protocol, SAP
Time Frame: Immediately following publication of primary project manuscript, or by 6 months after study completion, whichever is earlier.
Access Criteria: De-identified data will be made available through upload to the NITRIC Data Repository. As such, de-identified data will be publically available.